CLINICAL TRIAL: NCT02147392
Title: Assessment of [11C]ER-176 to Image Translocator Protein in Brain and Whole-Body of Healthy Subjects
Brief Title: Assessment of [11C]ER176 to Image Translocator Protein in Brain and Whole Body of Healthy People
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140117; 14-M-0117
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-01-26

CONDITIONS: Pharmacokinetics; Adult
Keywords: PET Imaging

INTERVENTIONS:
Drug: [11C]ER-176

SUMMARY:
Background:

- A protein called translocator protein may play a role in brain inflammation. Sometimes it is present at higher levels in the lungs than in the brain. Researchers want to see if a drug called [11C]ER176 can provide an image of this protein in the brain.

Objective:

- To test the ability of a drug to image a protein, and test how it is distributed in the body.

Eligibility:

- Healthy adults over age 18.

Design:

* Participants will be screened with medical history, physical exam, and blood and urine tests.
* Participants will have a PET scan of the brain using [11C]ER176. It will be injected through an intravenous tube into 1-2 arm veins. A tube may also be put into an artery at the wrist or elbow. Some participants will also have a lung scan.
* For the PET, participants will lie on a bed that slides in and out of a doughnut-shaped scanner. A plastic mask will be molded to their face and head. They may be wrapped with restraining sheets. The scan will last about 120 minutes. Blood may be taken during the scan.
* Blood and urine will be taken before and after the scan.
* During another visit, participants will have an MRI scan of the brain. Participants will lie on a table that slides in and out of a metal cylinder. A strong magnetic field and radio waves will take pictures of the brain. The scanner makes loud knocking noises. Participants will be given earplugs.
* Some participants will have only a whole-body PET scan using [11C]ER176.

DETAILED DESCRIPTION:
Objective

Translocator protein 18 kDa (TSPO) is highly expressed in activated microglia and reactive astrocytes in brain, and it may, thereby, be a useful biomarker of neuroinflammation. We developed [(11)C]PBR28 as a positron emission tomographic (PET) radioligand to bind to TSPO and measure its density. Although [(11)C]PBR28 has high in vivo specific signal, it is very sensitive to the high and low affinity states of TSPO, which are caused by the rs6971 single nucleotide polymorphism (SNP) in the fourth exon of the TSPO gene resulting in a nonconservative alanine-to-threonine substitution in position 147 of the encoded TSPO protein. This co-dominant mutation yields three genetic groups: HH, HL, and LL, where H is the high-affinity form and L is the low affinity form. The frequency of the L allele is approximately 30%; thus, the frequency of the LL homozygote is approximately 9%. The affinity of PBR28 to H and L forms differs about 50 fold; thus, LL carriers provide no measureable signal in brain from [(11)C]PBR28. We recently developed a new TSPO ligand ER176, the affinity of which differs by only 1.2 fold and therefore LL carriers should provide measureable brain uptake. The purpose of this study is to assess the potential of [(11)C]ER176 to image TSPO in brain, characterize its binding sensitivity in lung of healthy subjects from all three genetic groups, and to do whole-body imaging for biodistribution and estimation of radiation dosimetry in humans.

The present protocol will use a new PET ligand [(11)C]ER176 to 1) perform an initial whole-body scan after [(11)C]ER176 injection in a single healthy volunteer to confirm wide-spread distribution of radioactivity to different body organs (Phase 0); 2) perform kinetic brain scans in healthy volunteers of 3 different genotypes, with about half of these volunteers undergoing lung scans in the same session (Phase 1), and; 3) perform whole-body imaging in healthy volunteers (Phase 2).

This study will assess the relative robustness of absolute quantitation of TSPO in the brain of healthy subjects, using an arterial input function and pharmacokinetic modeling. In addition, lung imaging will provide in vivo binding sensitivity of [(11)C]ER176 to TSPO genotype. Furthermore, the whole-body imaging would estimate the radiation-absorbed doses for future use of [(11)C]ER176 in clinical studies.

Study Population

We will select up to 36 healthy adult female and male volunteers (age 18 and older) of 3 different TSPO genotypes for brain imaging, and up to 11 additional healthy volunteers for whole body dosimetry analysis.

Design

For absolute quantification of TSPO, up to 36 healthy controls (up to 12 each of three TSPO genotypes) will have brain PET imaging using [(11)C]ER176 and these subjects will have the arterial line and a brain MRI scan. In about half of those subjects from each genotype group, lungs will be scanned in the same session. For radiation dosimetry of [(11)C]ER176, up to 11 subjects will have whole-body PET imaging. These subjects will not have arterial line and MRI scans.

Outcome Measures

The primary outcome measures are: (a) To assess absolute quantitation of TSPO with [(11)C]ER176, we will determine the identifiability and time stability of distribution volume in the brain calculated with compartmental modeling. The difference in mean distribution volumes among subjects with different genotypes would be used to evaluate the genotype sensitivity of [(11)C]ER176. (b) To assess whole-body biodistribution and dosimetry of [(11)C]ER176 we will use the organ time-activity curves.

As secondary outcome measure, we will examine the effect of polymorphism on [(11)C]ER176 binding in lungs because lungs have much higher density of TSPO and may be more effective to show whether ER176 is sensitive to the SNP.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 or older.
* Able to give written informed consent.
* Healthy based on medical history, physical examination and laboratory testing.

EXCLUSION CRITERIA:

* Any current Axis I diagnosis.
* Clinically significant laboratory abnormalities.
* Positive test for HIV.
* Unable to have a MRI scan.
* History of neurologic illness or injury with the potential to affect study data interpretation.
* History of seizures, other than in childhood and related to fever.
* Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
* Inability to lie flat on camera bed for at least two hours.
* Pregnancy or breast feeding.
* Drug/alcohol abuse or dependence
* Current use of prescription or chronic (more than 3 continuous weeks) use of over-the-counter medications for pain, fever or other inflammation including prednisolone (Orapred), aspirin (Ecotrin), ibuprofen (Advil), and acetaminophen (Tylenol). The medications will be reviewed to see if subject can be in the study. If the subject is taking any medication that is not permitted, he/she may be in the study if the medication can be safely stopped for three weeks. The subject s primary care doctor will be contacted to stop a medication if necessary. A written permission will be obtained from the subject to contact his/her doctor.

Please note that exclusion criteria for the dosimetry subjects are the same reported above, except for MRI contraindications, because an MRI will not be performed in these subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05-14; Primary Completion 2016-06-16 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
The identifiability and time stability of distribution volume calculated with compartmental modeling and evaluate the genotype sensitivity of [11C]ER-176 | 1 year

SECONDARY OUTCOMES:
Whole-body biodistribution and dosimetry of [11C]ER-176. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Banati RB, Myers R, Kreutzberg GW. PK ('peripheral benzodiazepine')--binding sites in the CNS indicate early and discrete brain lesions: microautoradiographic detection of [3H]PK11195 binding to activated microglia. J Neurocytol. 1997 Feb;26(2):77-82. doi: 10.1023/a:1018567510105. PMID 9181482
- [Background] Banati RB, Newcombe J, Gunn RN, Cagnin A, Turkheimer F, Heppner F, Price G, Wegner F, Giovannoni G, Miller DH, Perkin GD, Smith T, Hewson AK, Bydder G, Kreutzberg GW, Jones T, Cuzner ML, Myers R. The peripheral benzodiazepine binding site in the brain in multiple sclerosis: quantitative in vivo imaging of microglia as a measure of disease activity. Brain. 2000 Nov;123 ( Pt 11):2321-37. doi: 10.1093/brain/123.11.2321. PMID 11050032
- [Background] Cagnin A, Brooks DJ, Kennedy AM, Gunn RN, Myers R, Turkheimer FE, Jones T, Banati RB. In-vivo measurement of activated microglia in dementia. Lancet. 2001 Aug 11;358(9280):461-7. doi: 10.1016/S0140-6736(01)05625-2. PMID 11513911
- [Derived] Kobayashi M, Jiang T, Telu S, Zoghbi SS, Gunn RN, Rabiner EA, Owen DR, Guo Q, Pike VW, Innis RB, Fujita M. 11C-DPA-713 has much greater specific binding to translocator protein 18 kDa (TSPO) in human brain than 11C-( R)-PK11195. J Cereb Blood Flow Metab. 2018 Mar;38(3):393-403. doi: 10.1177/0271678X17699223. Epub 2017 Mar 21. PMID 28322082